CLINICAL TRIAL: NCT03204942
Title: Comparison Between Dorsal Root Ganglion Thermal Radiofrequency Versus Pulsed Radiofrequency for the Management of Intractable Metastatic Pain in Thoracic Vertebral Body
Brief Title: Dorsal Root Ganglion Thermal Radiofrequency Versus Pulsed Radiofrequency for Metastatic Pain in Thoracic Vertebral Body
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Sherry N. Fanous, Principal Investigator, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CdGrPfMiPnB
Record Dates: First submitted 2017-06-11; First posted 2017-07-02 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Bone Neoplasm,Malignant Vertebral Column Thoracic Secondary
Keywords: Bone metastasis,Thoracic secondary, Cancer Pain,
MeSH Terms: conditions — Bone Neoplasms; Cancer Pain | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- PRF on DRG (Active Comparator): Patients will receive Pulsed Radiofrequency (PRF) on Dorsal root ganglion(DRG) of the selected metastatic painful dorsal vertebrae, with temperature 42°C for 480 sec.,2 active cycles per second of 20 milliseconds each , with a voltage output 40 to 60-V range, impedance ranges between 150 and 400 Ohms at all levels using Fluroscopic guidance (FG).
  Interventions: Device: PRF on DRG
- TRF on DRG (Active Comparator): Patients will receive Thermal Radiofrequency (TRF) on Dorsal root ganglion(DRG) of the selected metastatic painful dorsal vertebrae, with temperature 80°C for 90 sec.,2 cycles, using Fluoroscopic guidance (FG) .
  Interventions: Device: TRF on DRG
- Control group (Active Comparator): The control group will have identical needle placement and preparation like the 2 previous groups without the RF lesion, but with the injection of particulate Betamethasone steroids and local anesthetic on DRG of the selected metastatic painful dorsal vertebrae, using Fluoroscopic guidance (FG).
  Interventions: Drug: Corticosteroid injection

INTERVENTIONS:
Device: PRF on DRG — RF will be performed with the patient in a prone position with mild flexion of the spine. Fluoroscopy beam positioned in an antero-posterior direction. A 10 cm RF needle 20 G with a 10 mm active tip.The needle is inserted in a slightly medial-cephalad direction under the transverse processes, and using lateral fluoroscopic imaging, incrementally walking into the thoracic intervertebral foramen. So the location of the needle tip confirmed by sensory stimulation at 50 Hz. The point of maximum stimulation is at 0.5 V intensity and this is designated to be the location of the DRG. Slight redirection can be done to optimize the stimulation; injection of contrast reveals epidural uptake. After establishing the site for the RF, 1 ml 2% lidocaine should be injected through the needle.
  Arms: PRF on DRG
Device: TRF on DRG — Similar to the group of " PRF on DRG", but the types of the waves will be different as previously described
  Arms: TRF on DRG
Drug: Corticosteroid injection — Similar to the previous groups, but without applying any type of Radio-frequency but just injecting steroids and local anesthetics as previously described
  Arms: Control group

SUMMARY:
AIM OF THE WORK To evaluate the effectiveness and safety of Pulsed and Thermal Radiofrequency lesion of the dorsal root ganglion (RF-DRG) on a consecutive group of patients presenting with chronic thoracic pain due to vertebral bone metastasis.

DETAILED DESCRIPTION:
STUDY DESIGN This is a Prospective Randomized Controlled trial that will be conducted at the National Cancer Institute. All patients who are eligible for the study will be included and randomized into 3 equal groups.

PATIENTS AND METHODS After approval from the Ethics Committee at the National Cancer Institute, Cairo University, and obtaining written informed consent, eighty-one patients with thoracic segmental pain due to metastasis, unresponsive to conventional therapy and meeting the inclusion criteria will be randomly assigned to either one of the two types of treatment, PRF or TRF lesioning of the DRG or the control group. Patients will be carefully evaluated for neurologic deficits and side effects. Assessment of pain will be done at baseline then at 1, 3, 6 months after the procedure. Randomization will be done using randomized permuted block design. Randomization list will be generated through random.org online site.

Patients will be randomly assigned and divided into 3 equal comparable groups. Before the procedure, laboratory investigations, Dorsal X-ray, CT and MRI will be done. All Patients will be interviewed and examined by physicians trained in interventional pain management. Patients will be carefully assessed on physical exam for sensory, motor, or reflex deficit and carefully documented. Patients will be informed about the technique of the blocks, and written informed consents will be obtained.

The types of measures used to assess pain relief will include single rating scales; VAS, and multiple-dimension composite measures; Oswestry Low Back Pain Disability Questionnaire (ODI), The European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 and QLQ-BM22.

ELIGIBILITY:
Inclusion Criteria:

1. A greater than 6-month history of segmental pain of thoracic vertebral body metastasis origin.
2. Unsatisfactory pain control with oral pharmacotherapy including strong opioid with VAS >5 .
3. Absence of a chronic or progressive motor deficit.
4. Absence of significant sensory deficit.
5. No indication for percutaneous or open surgical intervention.
6. Magnetic resonance imaging and Computed Tomogrophy evidence of thoracic involvement.
7. ASA status of II to III .
8. Age > 18 .
9. Body mass index (BMI) :less than forty and more than twenty .
10. Informed consent

Exclusion Criteria:

1. Known sensitivity or contraindication to injected materials: local anesthetics.
2. History of psychological disorders.
3. Evidence of significant neurological deficit.
4. Inability to lie prone.
5. Local contraindication to procedure e.g. local sepsis at the site of intervention, coagulopathy.
6. Patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Na Fanous, M.Sc., Principal Investigator — National Cancer Institute, Egypt
Locations (1):
- Sherry Nabil Elia Fanous, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
All the data that will be found relevant to the primary and secondary outcome

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 140 patients were assessed for primary eligibility using Visual Analogue Scale(VAS).Of which81 only met the inclusion and exclusion criteria. Those 81 were assessed for final eligibility using MRI, CT and bone scan. 69 were included and12 were excluded before randomization due to4 died,4 declined to participate and4 had severe health deterioration
Groups:
- PRF on DRG: Patients will receive Pulsed Radiofrequency (PRF) on Dorsal root ganglion(DRG) of the selected metastatic painful dorsal vertebrae, with temperature 42°C for 480 sec.,2 active cycles per second of 20 milliseconds each , with a voltage output 40 to 60-V range, impedance ranges between 150 and 400 Ohms at all levels using Fluroscopic guidance(FG).
  PRF on DRG: RF will be performed with the patient in a prone position with mild flexion of the spine. Fluoroscopy beam positioned in an antero-posterior direction. A 10 cm RF needle 20 G with a 10 mm active tip.The needle is inserted in a slightly medial-cephalad direction under the transverse processes, and using lateral fluoroscopic imaging, incrementally walking into the thoracic intervertebral foramen. So the location of the needle tip confirmed by sensory stimulation at 50 Hz. The point of maximum stimulation is at 0.5 V intensity and this is designated to be the location of the DRG. Slight redirection can be done to optimize the st
Period: Overall Study
Arm/Group | PRF on DRG | TRF on DRG | Control Group
Started | 23 | 23 | 23
Completed | 23 | 23 | 23
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PRF on DRG: Patients received Pulsed Radiofrequency (PRF)on Dorsal root ganglion(DRG) of the selected metastatic painful dorsal vertebrae, with temperature 42°C for 480 sec.2 active cycles per second of 20 milliseconds each , with a voltage output 40-60-V ,impedance between 150-400 Ohms at all levels using Fluroscopic guidance. RF was performed with the patient in a prone position with mild flexion of the spine. Fluoroscopy beam positioned in an AP direction. A 10 cm RF needle 20 G with a 10 mm active tip.The needle was inserted in a slightly medial-cephalad direction under the transverse processes, and using lateral fluoroscopic imaging, incrementally walking into the thoracic intervertebral foramen. The location of the needle tip confirmed by sensory stimulation at 50 Hz. The point of maximum stimulation was at 0.5 V . injection of contrast reveals epidural uptake. After establishing the site for the RF, 1 ml 2% lidocaine was injected through the needle.
- TRF on DRG: Patients received Thermal Radiofrequency (TRF) on Dorsal root ganglion(DRG) of the selected metastatic painful dorsal vertebrae, with temperature 80°C for 90 sec.,2 cycles, using Fluoroscopic guidance (FG) .
  TRF on DRG: Similar to the group of " PRF on DRG", but the types of the waves was different as previously described
- Control Group: The control group had identical needle placement and preparation like the 2 previous groups without the RF lesion, but with the injection of particulate Betamethasone steroids and local anesthetic on DRG of the selected metastatic painful dorsal vertebrae, using Fluoroscopic guidance (FG).
  Corticosteroid injection: Similar to the previous groups, but without applying any type of Radio-frequency but just injecting steroids and local anesthetics as previously described
- Total: Total of all reporting groups
Arm/Group | PRF on DRG | TRF on DRG | Control Group | Total
Number analyzed (Participants) | 23 | 23 | 23 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.87 (10.55) | 55.78 (7.34) | 59.39 (13.72) | 55.8 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 13 | 41
  Male | 10 | 8 | 10 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 23 | 23 | 23 | 69
Region of Enrollment [Number; unit: participants]
  Egypt | 23 | 23 | 23 | 69
Interventional Level [Number; unit: participants]
  Dorsal vertebrae 3 | 1 | 1 | 2 | 4
  Dorsal vertebrae 4 | 1 | 4 | 2 | 7
  Dorsal vertebrae 5 | 4 | 6 | 4 | 14
  Dorsal vertebrae 6 | 5 | 9 | 3 | 17
  Dorsal vertebrae 7 | 4 | 7 | 3 | 14
  Dorsal vertebrae 8 | 2 | 8 | 4 | 14
  Dorsal vertebrae 9 | 4 | 4 | 6 | 14
  Dorsal vertebrae 10 | 7 | 1 | 4 | 12
  Dorsal vertebrae 11 | 3 | 0 | 1 | 4
  Dorsal vertebrae 12 | 6 | 0 | 4 | 10
Cancer Origin [Count of Participants; unit: Participants]
  Bladder | 1 | 0 | 1 | 2
  Breast | 10 | 12 | 12 | 34
  Chest Wall | 1 | 0 | 0 | 1
  Colon | 0 | 1 | 0 | 1
  Endometrial | 0 | 1 | 0 | 1
  Liver | 1 | 0 | 0 | 1
  Lung | 2 | 2 | 1 | 5
  Lymphoma non-Hodgikin | 0 | 1 | 1 | 2
  Lymphoma Hodgikin | 2 | 0 | 0 | 2
  Multiple Myeloma | 0 | 1 | 1 | 2
  Ovaries | 2 | 1 | 1 | 4
  Prostate | 3 | 3 | 4 | 10
  Stomach | 1 | 0 | 0 | 1
  Unknown | 0 | 1 | 2 | 3
Body Mass Index [Mean (Standard Deviation); unit: weight in kg divided by length in m2] | 27.54 (5.19) | 29.55 (6.08) | 28.50 (6.41) | 28.829 (5.78117)

OUTCOME MEASURES:

1. Primary Outcome: The European Organisation for Research and Treatment of Cancer (EORTC) Questionnaire to Measure Change in the Intensity of Pain QLQ-C30
Description: The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems e.g. a higher score in " Financial difficulties" represents a greater difficulty
Time Frame: Assessment done at 3 months after the procedure.
Population: At 3 months post intervention, there are changes in all groups in the Global health of the QLQ-C30 questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRF on DRG | TRF on DRG | Control Group
Number analyzed (Participants) | 23 | 23 | 23
score on a scale
  Global health status/QoL | 41.30 (9.56) | 51.08 (9.51) | 38.76 (12.47)
  Physical functioning | 42.48 (20.77) | 46.53 (19.10) | 54.96 (15.92)
  Role functioning | 59.16 (25.99) | 62.06 (21.89) | 65.67 (23.57)
  Emotional functioning | 33.42 (24.53) | 29.43 (22.83) | 50.09 (22.93)
  Cognitive functioning | 26.54 (25.44) | 30.16 (20.29) | 38.84 (18.62)
  Social functioning | 65.67 (22.47) | 62.05 (24.60) | 67.85 (25.28)
  Fatigue | 52.67 (16.51) | 49.27 (14.94) | 62.33 (13.72)
  Nausea and vomiting | 24.64 (23.49) | 28.26 (16.22) | 37.68 (23.69)
  Pain | 57.25 (18.01) | 45.64 (17.58) | 62.32 (14.40)
  Dyspnea | 31.87 (23.53) | 28.97 (23.15) | 43.47 (23.45)
  Insomnia | 52.17 (19.69) | 49.28 (24.37) | 55.07 (23.82)
  Appetite loss | 43.47 (27.42) | 37.67 (20.87) | 57.97 (25.08)
  Constipation | 30.43 (31.65) | 23.17 (21.16) | 34.77 (30.95)
  Diarrhea | 11.59 (19.09) | 11.58 (16.22) | 11.58 (16.22)
  Financial difficulties | 85.51 (24.26) | 82.61 (28.20) | 85.51 (26.26)

2. Primary Outcome: EORTC QLQ-BM22
Description: The scoring procedure for the QLQ-BM22 module is identical in principle to that for the function and symptom scales/items of the QLQ-C30. Each sub scale is then linearly converted to a score from 0 to 100. For the QLQ-BM22, a higher score indicates worse symptom burden for painful sites and pain characteristics, and better functioning for functional interference and psychosocial aspects. With regards to the positive phrasing of questions 21 and 22, the scoring must be reversed prior to statistical analysis. The item range for each scale/item is 3.
Time Frame: Assessment done at 3 months after the procedure.
Population: The QLQ-BM22 at 3 months post intervention there were changes in terms of Painful sites and Pain characteristics.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PRF on DRG: Patients received Pulsed Radiofrequency (PRF) on Dorsal root ganglion(DRG) of the selected metastatic painful dorsal vertebrae, with temperature 42°C for 480 sec.,2 active cycles per second of 20 milliseconds each , with a voltage output 40 to 60-V range, impedance ranges between 150 and 400 Ohms at all levels using Fluroscopic guidance (FG).
  A 10 cm RF needle 20 G with a 10 mm active tip.The needle was inserted in a slightly medial-cephalad direction under the transverse processes, and using lateral fluoroscopic imaging, incrementally walking into the thoracic intervertebral foramen. So the location of the needle tip confirmed by sensory stimulation at 50 Hz. The point of maximum stimulation was at 0.5 V intensity and this is designated to be the location of the DRG. After establishing the site for the RF, 1 ml 2% lidocaine was injected through the needle.
Arm/Group | PRF on DRG | TRF on DRG | Control Group
Number analyzed (Participants) | 23 | 23 | 23
score on a scale
  Painful Sites | 50.43 (16.80) | 35.07 (12.10) | 44.36 (16.65)
  Pain Characteristics | 41.54 (15.09) | 30.41 (13.90) | 34.75 (10.75)
  Functional Interference | 54.43 (22.62) | 52.08 (16.33) | 59.88 (14.64)
  Psychosocial Aspects | 51.90 (26.31) | 56.49 (20.42) | 51.41 (24.03)

3. Primary Outcome: Visual Analog Scale (VAS), to Evaluate Pain
Description: The VAS is a horizontal line,from 0 to 100 mm in length, anchored by word descriptors at each end such as "no pain" on the left and "severe pain" on the right. The patient marks on the line three pain ratings, corresponding to current, best and worst intensity of pain experienced over the past 24 hours.High VAS means worsening of pain. The average of the 3 ratings will be used to represent the patient's level of pain over the previous 24 hours. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.The VAS has consistently demonstrated sensitivity to changes in cancer pain associated with treatment or time ) and usually shows strong associations with other pain intensity ratings, it appears adequately valid and reliable as measures of pain intensity among the many different samples of persons with cancer
Time Frame: Assessment of pain done at 3 months after the procedure.
Population: Patients receiving PRF treatment changes in VAS% at 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRF on DRG | TRF on DRG | Control Group
Number analyzed (Participants) | 23 | 23 | 23
units on a scale | 68.57 (9.06) | 48.78 (9.55) | 66.17 (6.67)

4. Primary Outcome: Oswestry Low Back Pain Disability Questionnaire (ODI),
Description: ODI is a self-administered questionnaire divided into ten sections, each with six items designed to assess limitations of various activities of daily living. Each section is scored on a 0 to 5 scale, with 5 representing the greatest disability.If a patient marked more than one statement for a question, the highest scoring statement is recorded as the true indication of disability. The scores are assessed from 0% to 20% to indicate minimal disability, 20% to 40%, to indicate moderate disability, 40% to 60% to indicate severe disability, 60% to 80% to indicate crippled, and 80% to 100% to indicate bed bound or exaggerating their symptoms
Time Frame: Assessment of pain done at 3 months after the procedure.
Population: TRF group showed changes in pain and ODI% at 3 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- TRF on DRG: Patients received Thermal Radiofrequency (TRF) on Dorsal root ganglion(DRG) of the selected metastatic painful dorsal vertebrae, with temperature 80°C for 90 sec.,2 cycles, using Fluoroscopic guidance (FG) .
  TRF on DRG: Similar to the group of " PRF on DRG", but the types of the waveswas be different as previously described
Arm/Group | PRF on DRG | TRF on DRG | Control Group
Number analyzed (Participants) | 23 | 23 | 23
score on a scale | 62.52 (12.89) | 52.87 (11.86) | 61.61 (8.45)

5. Secondary Outcome: Number of Participants With Any Complications
Description: from either the technique as pneumothorax, Neurological defects, Dysthesia and hypoesthesia, anesthesia dolorosa and burning pain or local anesthetic complications.
Time Frame: Assessment done at 3 months after the procedure
Population: In the TRF group there were some changes
Measure: Number; unit: participants
Arm/Group | PRF on DRG | TRF on DRG | Control Group
Number analyzed (Participants) | 23 | 23 | 23
participants | 0 | 7 | 1

6. Secondary Outcome: To Measure Change in Analgesic Usage
Description: The change in the pre procedure use of different analgesics in comparison to 3 months later, using Analgesic Quantification Algorithm (AQA).0 No analgesic, 1 Non-opioid analgesics, 2 Weak opioids, 3 Strong opioids ≤75 mg OME per day, 4 Strong opioids >75-150 mg OME per day, 5 Strong opioids >150-300 mg OME per day, 6 Strong opioids >300-600 mg OME per day, 7 Strong opioids >600 mg OME per day.
Time Frame: Assessment was done before intervention and at at 3 months after the procedure.
Population: Opioid consumption varied in the 3 groups
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- TRF on DRG: Patients received Thermal Radiofrequency (TRF) on Dorsal root ganglion(DRG) of the selected metastatic painful dorsal vertebrae, with temperature 80°C for 90 sec.,2 cycles, using Fluoroscopic guidance (FG) .
  TRF on DRG: Similar to the group of " PRF on DRG", but the types of the waveswas different as previously described
Arm/Group | PRF on DRG | TRF on DRG | Control Group
Number analyzed (Participants) | 23 | 23 | 23
score on a scale
  Before intervention | 4.30 (1.11) | 4.57 (1.12) | 3.87 (0.87)
  After 3 months | 3.43 (1.12) | 2.70 (1.26) | 3.52 (0.95)

7. Secondary Outcome: Patients' Satisfaction, Descriptive Scale
Description: Patients' satisfaction with analgesia through a phone call on 5-level likert scale, (not satisfied at all, only slightly satisfied, somewhat or partly satisfied, very satisfied, perfectly satisfied )
Time Frame: a week after procedure
Population: improvement at 5-level Likert Scale was measured in all groups.
Measure: Count of Participants; unit: Participants
Arm/Group | PRF on DRG | TRF on DRG | Control Group
Number analyzed (Participants) | 23 | 23 | 23
Participants
  Very satisfied, perfectly satisfied | 1 | 16 | 0
  Somewhat or partly satisfied | 5 | 2 | 6
  Neutral | 9 | 4 | 4
  Only slightly satisfied | 7 | 1 | 13
  Not satisfied at all | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the study course ( 3 months)
Description: Adverse event were collected just post procedure by clinical examination then at 3 months post procedure.
Arm/Group | PRF on DRG | TRF on DRG | Control Group
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 7/23 | 1/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRF on DRG (N=23) | TRF on DRG (N=23) | Control Group (N=23)
Neuritis (Nervous system disorders) | 0 | 4 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Numbness (Nervous system disorders) | 0 | 2 | 0
Dysethsia (Nervous system disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT03204942/Prot_SAP_000.pdf